CLINICAL TRIAL: NCT00959751
Title: Phase 2 Study of the Safety and Effectiveness of a Single Oral Dose of NXN-188 for the Treatment of Moderate to Severe Migraine Headache Without Aura
Brief Title: Study of the Safety and Effectiveness of NXN-188 for the Treatment of Migraine Headache Without Aura
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NeurAxon Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NXN-188-204
Record Dates: First submitted 2009-08-14; First posted 2009-08-17 (Estimated); Results first posted 2014-07-11 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-07

CONDITIONS: Migraine Without Aura
Keywords: migraine
MeSH Terms: conditions — Migraine without Aura; Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NXN-188 600 mg (Experimental): 3 x 200 mg capsules, PRN
  Interventions: Drug: NXN-188
- Placebo (Placebo Comparator): 3 x 0 mg capsules, PRN
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NXN-188 — 200 mg capsules, 600 mg, PRN
  Other Names: NXN-188 dihydrochloride
  Arms: NXN-188 600 mg
Drug: Placebo — 200 mg capsules with no active ingredient designed to match the NXN-188 capsules
  Arms: Placebo

SUMMARY:
This is a a multi-center, randomized, double-blind, parallel group, and placebo controlled, two-arm study of a single oral dose of NXN-188 for the treatment of acute migraine headache without aura. Up to 120 migraineurs will be enrolled. Approximately 60 subjects having a headache history of migraine without aura will complete each of the two treatment arms to evaluate NXN-188 600 mg or placebo.

DETAILED DESCRIPTION:
After study eligibility was confirmed and all screening procedures completed, subjects were randomized at Visit 1 to receive either NXN-188 600 mg or placebo in a 1:1 ratio. Study drug and diaries were dispensed, and subjects were instructed regarding when to dose with study drug. Subjects were also trained regarding the Interactive Voice Response System (IVRS), and made familiar with the study diary and the completion of study diary assessments. Subjects left the clinic to self-administer treatment as an outpatient at the onset of a moderate to severe migraine headache without aura (as rated on a 4-point categorical scale). Dosing with study drug was to take place within 42 days from Randomization (Visit 1). The subject contacted the investigatorI or designee at 14 and 28 days after Randomization if they had not yet treated a migraine headache without aura in order to receive verbal permission from the site personnel to continue in the study as appropriate. If the subject had not treated a migraine headache within 42 days of Visit 1, the subject did not take study drug and returned all materials, including the unused study drug, to the study site. If the subject experienced a qualifying migraine without aura during the treatment period, (s)he recorded headache symptoms in the study diary when first noticed (and menstrual cycle status [female subjects only]). If the subject met dosing requirements as outlined in the protocol, they dosed with the study drug, called the IVRS to report dosing, recorded all assessments and adverse events (AEs) and contacted the study center to schedule a post treatment visit (Visit 2) within 6 days (± 2 days) of treatment. If study drug resulted in insufficient relief at 2 hours p.a., subjects were permitted to use the non-triptan rescue medication recommended by the PI at Visit 1. Within 6 days (± 2 days) of treatment, the subject returned to the study center for Visit 2. The subject had a brief physical examination, a 12-lead electrocardiogram (ECG), and had samples taken for clinical laboratory tests, including a serum pregnancy test for all females. Concomitant medications taken and adverse events (AEs) experienced from time of dosing to Visit 2 were reported to site personnel and recorded. Study diaries were reviewed and information recorded. Discontinuing subjects returned unused study drug and study material. One safety follow-up telephone contact was made within 15 days (± 2 days) post treatment. For those subjects not meeting the Treatment/Enrollment criteria by Day 42 (i.e., not experiencing a qualifying headache) and for other subjects discontinuing the study protocol post Randomization (Visit 1), a second visit, Visit 2, was required and subjects underwent a brief physical examination, had vital signs and ECGs performed, samples collected for clinical labs, concomitant medications and AEs reviewed, and returned all study drug and study materials.

ELIGIBILITY:
Inclusion Criteria:

1. Meets the following criteria for migraine headache without aura: Previously diagnosed with a history of migraine headaches; Headache has at least two (2) of the following characteristics: Unilateral location; Pulsating quality; Moderate or severe pain intensity; Aggravation by routine physical activity such as walking or climbing stairs; During headache, has at least one of the following characteristics: Nausea and/or vomiting; Photophobia and/or phonophobia;Not attributable to another disorder
2. Headache frequency of at least 2 migraine attacks per month for the past 3 months but not more than 8 migraines in any 30 day period. Each migraine attack should last at least 4 hours (without treatment) and not longer than 72 hours.
3. At the time of the study migraine, prior to dosing with study medication, the headache severity, as judged and documented by the subject, is either moderate or severe
4. BMI within the range of 18 to 35
5. Good general health as determined by the medical history, physical exam, clinical laboratory tests, vital signs and electrocardiogram. ALT cannot be above 1.5x upper limit of normal; creatinine and urea must be within normal limits
6. Speak, read, and understand English or French, sufficiently to understand the nature of the study, to provide written informed consent, and complete all study assessments.
7. Willing and able to comply with all testing requirements defined in the protocol
8. Females will avoid pregnancy at least 10 days before randomization, during the study and up until 3 months after treatment
9. All subjects/partners must use a double-barrier method of birth control during the study and for 3 months after dosing (female subjects who have had a tubal ligation > 1 year or who are post menopausal or post hysterectomy > 1 year and male subjects who are surgically sterile are exempted from this inclusion criteria.

Exclusion Criteria:

A diagnosis of headaches that is not consistent with migraine without aura as defined in the inclusion criteria. Subjects with a history of migraine with aura are excluded.

1. Presence of any risk factors that would preclude the use of triptans: Uncontrolled hypertension; Ischemic heart disease; Prinzmetal angina; Cardiac arrhythmias; Multiple risk factors for ischemic atherosclerotic vascular disease; Primary vasculopathies; Basilar and hemiplegic migraine
2. Known allergy or hypersensitivity to triptans or history of any serious side effect with a triptan which would preclude further dosing with a triptan
3. Presence of any clinically significant condition that would preclude study participation, as evaluated by the investigator
4. Pregnant or lactating
5. History of significant neurological, hepatic, renal, endocrine, cardiovascular, gastrointestinal, pulmonary, rheumatologic, autoimmune, or metabolic disease
6. Any use (within 30 days of randomization) of migraine prevention medication including: Valproate (Depakote), topiramate (Topamax), cyproheptadine (Periactin), montelukast (Singulair), or botulinum toxin, type A (Botox); Cardiovascular drugs (acceptable if reason for use is for treatment of cardiovascular disease and the subject has been on a stable dose; MAOIs within 30 days of randomization
7. Initiation of therapy with SSRIs or SNRIs for depression or other approved indication within 90 days of randomization (subjects on stable dose for >3 months for treatment of depression or other approved indication may be included)
8. Are known to or suspected to be currently abusing alcohol or drugs, or have a history (within the past 12 months) of active alcohol or drug abuse
9. Participation in another drug or biologic study within 30 days of randomization into this study or during participation in this study
10. Subjects unable or unwilling, in the opinion of the Investigator, to comply with all study procedures and cooperate fully with study center staff

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2009-07; Primary Completion 2010-02 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guy Boudreau, MD, Principal Investigator — Hopital Notre-Dame Du Chum, Montreal
Locations (4):
- United States (4):
  - Comprehensive Neuroscience, Inc., St. Petersburg, Florida
  - Comprehensive NeuroScience, Inc. Atlanta, Atlanta, Georgia
  - Elkind Headache Center, Mount Vernon, New York
  - Lifetree Clinical Research, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study Period - 6 months. First subject screened 28 July 2009, Last subject completed the study 9 February 2010.
Groups:
- Placebo: 3 x capsules, PRN
Period: Overall Study
Arm/Group | Placebo | NXN-188 600 mg
Started | 97 | 98
Completed | 88 | 86
Not Completed | 9 | 12
Not completed — Lost to Follow-up | 2 | 3
Not completed — Consent Withdrawn | 0 | 1
Not completed — Non-compliance to Study Procedures | 0 | 1
Not completed — No migraine headache without aura | 7 | 7

BASELINE CHARACTERISTICS:
Population: Of the 195 subjects randomized, 174 subjects received study drug: the 174 subjects constitute the Safety Population.
Groups:
- NXN-188: 3 x 200 mg capsules
- Placebo: 3 x 0 mg capsules
- Total: Total of all reporting groups
Arm/Group | NXN-188 | Placebo | Total
Number analyzed (Participants) | 86 | 88 | 174
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.2 (12.34) | 38.4 (12.63) | 39.3 (12.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 74 | 140
  Male | 20 | 14 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 13 | 34
  Not Hispanic or Latino | 65 | 75 | 140
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 19 | 32
  White | 72 | 66 | 138
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 74.94 (14.695) | 74.74 (17.066) | 74.84 (15.893)
Height [Mean (Standard Deviation); unit: cm] | 168.33 (8.502) | 165.91 (9.960) | 167.10 (9.321)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.2 (4.09) | 27.2 (5.28) | 26.7 (4.74)
Type of Migraine [Number; unit: Participants] — Subjects are counted once within each type where at least one migraine is recorded.
  Participants
    Without Aura | 86 | 88 | 174
    With Aura | 0 | 0 | 0
Number of Previous Migraines [Mean (Standard Deviation); unit: migraine episodes] — Previous Migraines for each subject was based on the total number of migraine entries reported on the Migraine History CRF
  migraine episodes | 1.1 (0.30) | 1.1 (0.23) | 1.1 (0.27)

OUTCOME MEASURES:

1. Primary Outcome: Headache Relief (Modified LOCF - Efficacy Evaluable Analysis Set)
Description: Headache relief at 2 hours post administration defined as reduction from Baseline moderate or severe score to mild or none.
Time Frame: 2 hours
Population: Modified LOCF - Efficacy Evaluable Analysis Set
Measure: Number; unit: Participants
Arm/Group | NXN-188 600 mg | Placebo
Number analyzed (Participants) | 80 | 79
Participants | 42 | 30

2. Secondary Outcome: Headache Relief Based on a 2-Point Reduction From Baseline (Modified LOCF - Efficacy Evaluable Analysis Set)
Description: The Headache Severity Score (HSS) assessment was recorded in the diary by the subject and used the following categories: 0 = no pain; 1 = mild pain; 2 = moderate pain; and, 3 = severe pain
Time Frame: 72 hours
Measure: Number; unit: Participants
Arm/Group | NXN-188 600 mg | Placebo
Number analyzed (Participants) | 80 | 79
Participants
  Headache Relief - 2 hours | 28 | 17
  Headache Relief - 4 hours | 45 | 26
  Headache Relief - 24 hours | 59 | 42
  Headache Relief - 72 hours | 54 | 47

3. Secondary Outcome: Headache Relief Based on a 1-Point Reduction From Baseline (Modified LOCF - Efficacy Evaluable Analysis Set)
Description: as for outcome 2
Time Frame: 72 hours
Measure: Number; unit: Participants
Arm/Group | NXN-188 600 mg | Placebo
Number analyzed (Participants) | 80 | 79
Participants
  Headache Relief - 2 hours | 52 | 40
  Headache Relief - 4 hours | 63 | 46
  Headache Relief - 24 hours | 64 | 52
  Headache Relief - 72 hours | 62 | 52

4. Secondary Outcome: Complete Headache Relief (Efficacy Evaluable Analysis Set)
Time Frame: 72 hours
Measure: Number; unit: Participants
Arm/Group | NXN-188 600 mg | Placebo
Number analyzed (Participants) | 80 | 79
Participants
  Complete Headache Relief - 2 hours | 19 | 9
  Complete Headache Relief - 4 hours | 35 | 19
  Complete Headache Relief - 24 hours | 56 | 36
  Complete Headache Relief - 72 hours | 54 | 43

5. Primary Outcome: Headache Recurrence (Modified LOCF - Efficacy Evaluable Analysis Set)
Description: Headache recurrence is defined as any subject that experiences headache relief at the given time point (i.e., 2 hours or 4 hours), who did not use rescue medication and who experienced a worsening of their headache to moderate or severe within 24 hours following study drug administration. The denominator is the number of subjects who experienced headache relief at 2 hours/4 hours.
Time Frame: 4 hours
Population: 30 and 42 placebo and NXN-188 subjects, respectivley, experienced headache relief at 2 hours. 41 and 55 placebo and NXN-188 subjects, respectively, experienced headache relief at 4 hours.
Measure: Number; unit: Participants
Arm/Group | NXN-188 600 mg | Placebo
Number analyzed (Participants) | 80 | 79
Participants
  Headache Recurrence - 2 hours | 3 | 6
  Headache Recurrence - 4 hours | 2 | 4

6. Secondary Outcome: Time (Hours) to First Use of Rescue Medication (Full Analysis Set)
Description: Subjects who do not require rescue medication are censored at the time of their last diary assessment completed up to 24 hours following study drug administration.
Time Frame: 24 Hours
Population: Full Analysis Set includes all subjects in the Safety Population who had at least one post-dose observation for headache severity recorded in his or her diary.
Measure: Median (95% Confidence Interval); unit: Participants who required rescue
Arm/Group | NXN-188 600 mg | Placebo
Number analyzed (Participants) | 86 | 88
Participants who required rescue | NA [NA to NA] — Median times not estimable by Kaplan-Meier because too few subjects required rescue medication within 25 hrs | NA [19.6 to NA] — Median times not estimable by Kaplan-Meier because too few subjects required rescue medication within 24 hrs

7. Secondary Outcome: Overall Evaluation of Study Medication at 24 Hours Post Administration (Full Analysis Set)
Description: Overall evaluation of the study drug was measured with a 4-point scale at 24 hours and used the following categories: 1 = Poor; 2 = Moderate; 3 = Good; and,4 = Excellent
Time Frame: 24 hours
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | NXN-188 600 mg | Placebo
Number analyzed (Participants) | 86 | 88
Participants
  1 = Poor | 20 | 37
  2 = Moderate | 22 | 19
  3 = Good | 26 | 21
  4 = Excellent | 18 | 11

8. Post Hoc Outcome: Sustained Complete Headache Relief (Efficacy Evaluable Analysis Set)
Description: Exploratory Post-hoc Analysis: Sustained complete headache relief is defined as a reduction in headache severity from moderate or severe to absent over all indicated time points.
Time Frame: 2 - 48 hours
Population: Efficacy Evaluable Analysis Set includes all subjects in the Full Analysis Set with an observed or imputed HSS (using rules predefined in the Statistical Analysis Plan [SAP]) at both the 2-hour time point and the 4-hour time point when using the modified LOCF approach
Measure: Number; unit: Participants
Arm/Group | NXN-188 600 mg | Placebo
Number analyzed (Participants) | 80 | 79
Participants
  2-24 hours | 17 | 8
  4-24 hours | 32 | 18
  2-48 hours | 16 | 8
  4-48 hours | 29 | 18

ADVERSE EVENTS:
Time Frame: Adverse event data were collected throughout the study beginning with the dosing of study drug and ending 15 days (± 2 days) p.a.
Description: All AE summaries were restricted to TEAEs, which were defined as those AEs that occurred after dosing and those existing AEs that worsened during the study.
Arm/Group | NXN-188 600 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/86 | 1/88
Other Adverse Events (participants affected / at risk) | 17/86 | 13/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NXN-188 600 mg (N=86) | Placebo (N=88)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NXN-188 600 mg (N=86) | Placebo (N=88)
Nausea (Gastrointestinal disorders) | 4 (4) | 7 (7)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 5 (8) | 3 (3)
Somnolence (Nervous system disorders) | 1 (1) | 2 (2)
Chills (General disorders) | 2 (2) | 0 (0)
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Proteinuria (Renal and urinary disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor may request Investigator or Institution not to publish or disclose information related to the clinical study.